CLINICAL TRIAL: NCT00067184
Title: Methadone, Buprenorphine and Fetal Development
Brief Title: Fetal Neurobehavioral Development in Methadone Maintained Pregnancies
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: HBV98112004; R01DA019934 (NIH); DPMCDA
Record Dates: First submitted 2003-08-12; First posted 2003-08-13 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Opioid-Related Disorders
Keywords: methadone; fetus
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Toitu 320/325 — Fetal monitor

SUMMARY:
The purpose of this study is to examine differences in fetal neurobehavior at peak (2 hours after oral dose) vs. trough (2 hours before oral dose) maternal plasma methadone levels.

DETAILED DESCRIPTION:
This study will examine differences in fetal neurobehavior at peak (2 hours after oral dose) vs. trough (2 hours before oral dose) plasma methadone levels. Anecdotal clinical observations suggest that fetal activity is increased at trough methadone levels and decreased at peak methadone levels, yet the investigators do not understand how in utero methadone exposure affects fetal neurobehavioral state development.

ELIGIBILITY:
Actively enrolled pregnant patients in CAP SA treatment.

Inclusion Criteria:

* Maternal age 18-40 years
* Single intrauterine fetus
* Estimated gestational age of 32 weeks
* DSMIV criteria for opioid dependence according to e-module of the SCID
* Daily methadone maintenance at a stable dose for greater than a week

Exclusion Criteria:

* Concurrent DSMIV axis I diagnosis that would preclude informed consent procedures (i.e., schizophrenia, major depression) or confound study outcomes (e.g., Alcohol Dependence)
* Presence of a serious medical or psychiatric illness requiring chronic medication or other intervention (i.e., HIV infection) that may confound data interpretation
* Evidence of preterm labor
* Evidence of prescription drug use (e.g., antidepressants, tranquilizers)
* Presence of major congenital fetal malformation
* Recent use (last month) of other illicit drugs (e.g., cocaine, marijuana) based on self report or positive on-Trak urine drug toxicology at time of actograph sessions
* Split methadone dosing schedule

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Methadone exposed pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2002-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
fetal heart rate | 120 minutes
fetal movement | 120 minutes

SECONDARY OUTCOMES:
neonatal abstinence syndrome | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M. Jansson, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Addiction and Pregnancy, Baltimore, Maryland, United States

REFERENCES:
- [Result] Jansson LM, Dipietro J, Elko A. Fetal response to maternal methadone administration. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 1):611-7. doi: 10.1016/j.ajog.2005.02.075. PMID 16150250